CLINICAL TRIAL: NCT05906914
Title: A Monocenter Prospective Single Arm Study of Cladribine Plus Homoharringtonine and Cytarabine Regimen (CHA) for Induced Therapy in Adults de Novo Acute Myeloid Leukemia (Non-M3)
Brief Title: Cladribine Plus Homoharringtonine and Cytarabine Regimen (CHA) for de Novo Acute Myeloid Leukemia
Acronym: CHA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20220027C-R2
Record Dates: First submitted 2023-05-14; First posted 2023-06-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cladribine; Homoharringtonine; Cytarabine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Group (Experimental): Intervention: CHA
  Interventions: Drug: cladribine + homoharringtonine + cytarabine

INTERVENTIONS:
Drug: cladribine + homoharringtonine + cytarabine — CHA Protocol: cladribine (5mg/m2, d1-3) + homoharringtonine (2mg/m2, d1-5) + cytarabine (100mg/m2 d1-7).
  Other Names: Cladribine Injection; Cytarabine for injection; Homoharringtonine Injection

SUMMARY:
The goal of this clinical trial is to evaluate the response and safety of Cladribine plus Homoharringtonine and Cytarabine regimen (CHA) protocol in de novo acute myeloid leukemia with age <60y. This is a prospective, single-armed mono-center based investigator-initiated trial. About 30 patients who meet the enrollment criteria with be treated with CHA as induction chemotherapy. The complete response rate, survival rate, recurrence rate, and treatment-related mortality with be observed.

DETAILED DESCRIPTION:
In this study, a new chemotherapy regimen named CHA which composed of cladribine, homoharringtonine and cytarabine, was proposed for the induced remission treatment of adult acute myeloid leukemia, and the efficacy and safety of this regimen were evaluated. Enrolled patients will receive cladribine (5mg/m2, d1-3) + homoharringtonine (2mg/m2, d1-5) + cytarabine (100mg/m2, d1-7). If more than partial remission is achieved in the first course, a course of CHA regimen is repeated. If the first course of treatment did not achieve a partial response, or the second course of treatment did not achieve a complete response, the patient was withdrawn from the clinical study. Transplantation was stratification according to the prognostic risk stratification. Patients with favourable risk received 3 cycles of high-dose intravenous cytarabine (1-3g/m2, Q12H d1-3). Or 3 cycles of medium dose cytarabine (1.0g/m2, Q12H d1-3) combined with idarubicin (10mg/m2, d1-3) or etoposide (100mg, d1-3). Patients with intermediate risk who achieve minimal residual disease (MRD) negative in the first or second cycle can receive high-dose or intermediate-dose cytarabine chemotherapy, otherwise allogeneic hematopoietic stem cell transplantation (HSCT) is recommended. Patients with high risk are advised to receive allogeneic HSCT, or receive high-dose or intermediate-dose cytarabine.Bone marrow samples were collected at enrollment for bone marrow cytology, flow cytometry and next-generation sequencing. The probes for targeted sequencing covered exons and selected introns of 88 myeloid leukaemia-related genes for next-generation sequencing. Bone marrow was collected on day 28 after each treatment cycle, including bone marrow cytology and measurable residual disease (MRD) assessments, for response assessment.The response assessment was evaluated according to the Revised Recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. The primary study endpoint was the composite complete remission (CR) rate (CR and CR with incomplete hematology recovery, CRi), assessed in all treated populations according to the Revised Recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. The secondary endpoints were minimal residual disease in bone marrow measured by flow cytometry after one cycle of induction therapy, as well as overall survival (OS), event-free survival, and adverse events, assessed in all treated populations.

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18 to 59 years old, gender is not limited, race is not limited.
2. Diagnosed as acute myeloid leukemia (AML) according to the diagnostic criteria of the World Health Organization (WHO) in 2016.
3. No previous anti-acute leukemia therapy (including demethylation drugs for leukemia or myelodysplastic syndrome (MDS), except hydroxyurea and leukocytosis).
4. Physical status <= 2 according to eastern tumor cooperation group (ECOG).
5. Within 21 days before random grouping and at baseline, biochemical indicators must be within the following limits: Glutamic pyruvic transaminase (ALT) and glutamic oxaloacetic transaminase (AST) <= 3 × normal upper limit (ULN); total bilirubin <= 3 × ULN; serum creatinine <= 2 × ULN or serum creatinine clearance rate (CrCl)>= 40mL/min.
6. The left ventricular ejection fraction| (LVEF) measured by echocardiography was in the normal range (LVEF > 50%).
7. Each patient (or his or her legal representative) must sign an informed consent form (ICF), indicating that he / she understands the purpose and procedures of the study and is willing to participate in the study.

Exclusion Criteria:

1. Diagnosed or receiving treatment for other malignant tumors other than AML that are or are in need of treatment in the near future.
2. Acute promyelocytic leukemia, myeloid sarcomas, accelerated and acute transformation of chronic myeloid leukemia.
3. Patients with severe liver and kidney function, cardiopulmonary insufficiency.
4. Uncontrolled or severe infection.
5. Mental illness that may prevent subjects from completing treatment or informed consent.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate | At the end of Cycle 1 (each cycle is 28 days)
  no signs of leukemia after treatment, fewer than 5% blasts in the BM, absolute neutrophil count (ANC) ≥ 1.0×109/L and platelet count ≥ 100×109/L and absence of the extramedullary tumor
Overall Survival Rate | 2 years since enrollment
  the ratio of cases alive to total enrolled cases within 2 years since enrollment
Disease-free Survival Rate | 2 years since enrollment
  the ratio of cases with leukemia complete remission to the total enrolled cases within 2 years since enrollment

SECONDARY OUTCOMES:
Recurrence Rate | 2 years since enrollment
  the ratio of cases with leukemia relapse to the total enrolled cases within 2 years since enrollment
Treatment-related mortality | 30 days since treatment
  the ratio of cases who died within 30 days since treatment to total enrolled cases

CONTACTS AND LOCATIONS:
Overall Officials: Jie Sun, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China